CLINICAL TRIAL: NCT03809026
Title: The Potential of Sperm Retrieved by Micro-TESE to Fertilize Vitrified/Warmed Oocytes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Jens Fedder, Professor, MD, PhD, Odense University Hospital
Other Study IDs: Lab.Reprod.Biol. - Odense.03
Record Dates: First submitted 2019-01-16; First posted 2019-01-18 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-11

CONDITIONS: Azoospermia, Nonobstructive
Keywords: Azoospermia; micro-TESE; Klinefelter's syndrome; Cryptorchidism; Vitrified oocytes
MeSH Terms: conditions — Azoospermia, Nonobstructive; Azoospermia; Klinefelter Syndrome; Cryptorchidism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: Couples where the men have Klinefelter's syndrome, maturation stop in the spermatogenesis or failed retrieval of testicular sperm by conventional techniques with needle or TruCut, and where testicular sperm could be obtained by micro-TESE.
- Control group: Couples as in the study group, but where testicular sperm could not be obtained by micro-TESE. The oocytes therefore must be fertilized using donor sperm.

SUMMARY:
Couples referred for microdissection-TESE (m-TESE) due to Klinefelter's syndrome, maturation stop in the spermatogenesis, or failed retrieval of testicular spermatozoa by conventional techniques with needle or TruCut are included. The women are stimulated with FSH in IVF protocols and the aspirated oocytes vitrified with usual applied techniques. Fresh sperm retrieved by micro-TESE are used for fertilization of the warmed oocytes. when it is not possible to obtain testicular sperm, the couples are offered fertilization with warmed oocytes.

Fertilization, cleavage, implantation and pregnancy rates using sperm from the patients versus from sperm donors will be compared.

ELIGIBILITY:
Inclusion Criteria:

Couples referred for micro-TESE

Exclusion Criteria:

None

Ages: 18 Years to 100 Years | Sex: Male
Age Groups: Adult, Older Adult
Gender Based: Yes — Actually we treat infertile couples with a man and a woman, but the variable originates from the man.
Study Population: Men referred to micro-TESE due to Klinefelter's syndrome, maturation stop in the spermatogenesis, or failed sperm retrieval using conventional needles or TruCut.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-09-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Cleavage rate | six years
  Measurement of % of cleavage among the warmed oocytes
Pregnancy rate | six years
  Measurement of serum-hCG and ultrasonography at gestation age week 7
Fertilization rate | six years
  Measurement of % of fertilization among the warmed oocytes

SECONDARY OUTCOMES:
Implantation rate | six years
  Measurement of the % of transferred embryos implanting into the uterus

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Centre of Andrology & Fertility Clinic, Department D, Odense University Hospital, Odense
  - Centre of Andrology & Fertility Clinic, Odense University Hospital, Odense

IPD SHARING:
Plan to Share IPD: Undecided